CLINICAL TRIAL: NCT07116512
Title: Randomized, Non-blinded, Two-way Crossover Study to Assess Bioequivalence Between Finerenone Study Intervention A (Test) and Study Intervention B (Reference) in Healthy Male Adult Participants
Brief Title: A Study to Compare How Much of the Study Treatment Finerenone Gets Into the Blood When the Same Amount is Taken in One and in Two Tablets of Different Strengths in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 22292; 2022-502385-24 (Other: CTIS (EU))
Record Dates: First submitted 2025-08-06; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2024-07

CONDITIONS: Heart Failure With Left Ventricular Ejection Fraction Greater Than or Equal to 40 Per Cent; Healthy Volunteers
MeSH Terms: interventions — finerenone

STUDY DESIGN:
Intervention Model Description: Two-way crossover design
Masking Description: The study was performed in a non-blinded design (i.e., investigator and participants were not blinded).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- finerenone sequences: intervention A_intervention B (Experimental): Participants received intervention A first, with a washout period of at least 72 hours, participants then received intervention B
  Interventions: Drug: Finerenone (BAY94-8862): intervention A; Drug: Finerenone (BAY94-8862): intervention B
- finerenone sequences: intervention B_intervention A (Experimental): Participants received intervention B first, with a washout period of at least 72 hours, participants then received intervention A
  Interventions: Drug: Finerenone (BAY94-8862): intervention A; Drug: Finerenone (BAY94-8862): intervention B

INTERVENTIONS:
Drug: Finerenone (BAY94-8862): intervention A — Study intervention A: one tablet of dose strength 1 one tablet of dose strength 1 = two tablets of dose strength 2
Drug: Finerenone (BAY94-8862): intervention B — Study intervention B: two tablets of dose strength 2 two tablets of dose strength 2 = one tablet of dose strength 1

SUMMARY:
In this bioequivalence study, healthy male participants took the study treatment finerenone in the form of one and two tablets of different strengths by mouth. "Bioequivalence" means that the researchers want to show similar blood levels of finerenone in the participants when they take the one tablet form of finerenone compared to the two tablets form. This study helped researchers learn more about a new finerenone tablet with higher strength, which is being developed to treat people who have heart failure (HF) with left ventricular ejection fraction (LVEF) ≥ 40%.

HF with LVEF ≥ 40% is a condition which occurs when the left side of the heart does not pump blood out to the body as well as it should. Over time, the body does not get the amount of oxygen it needs. This can lead to shortness of breath and tiredness, making it harder for people to do their daily tasks.

Finerenone works by blocking a certain protein, called mineralocorticoid receptor. By doing this, finerenone reduces damage to kidneys, heart and blood vessels. It is available and approved for doctors to prescribe to people with chronic kidney disease together with type 2 diabetes.

The main objective of this study was to compare how much finerenone gets into the blood when the participants took the same amount of finerenone in the form of one and two tablets of different strengths by mouth.

Another objective of this study was to learn the degree to which medical problems that might be caused by finerenone can be tolerated (also called "tolerability") by the participants. These medical problems were also known as "adverse events". Doctors kept track of all adverse events that happened in the study, even if they did not think they might be related to the study treatments.

The study was conducted in a single-center, randomized, non-blinded, two-way crossover design in healthy male participants aged 18 to 55 years.

"Single-center" means at one research center or one hospital. "Randomized" means that the study participants were randomly (by chance) assigned to one of two sequences of treatments. "Non-blinded" means that both the participants and the study doctors and their team know what the participants will take. In a "two-way crossover" study, all the participants take all of the treatments, but in a different order. Each participant was in the study for approximately 4-6 weeks including a stay in the center for up to 6 days with 5 overnight stays.

In this study, each participant took finerenone twice by mouth on an empty stomach. They took finerenone in the form of one and two tablets of different strengths. The tablet form that was taken first depended on the treatment sequence to which the participants were assigned. There was a period of 3 days between the intake of the tablets.

Each participant served as his/her own control. This means that researchers made comparisons between the two tablet forms of finerenone within the same participant.

During the study, the doctors and their study team took blood and urine samples, did physical examinations, performed ECG and checked vital signs such as blood pressure, heart rate and body temperature.

Participants of this study were healthy and had no benefit from taking the study treatment finerenone. However, the study provided information on how to use the new tablet form of finerenone to treat patients with HF with LVEF ≥ 40% Specific measures had been put in place to counter and minimize the risks related to the conduct of this study. Information on safety of finerenone was already available from previous studies. Monitoring procedures, limitation of given doses and exclusion criteria had been defined. Blood samples were taken via an indwelling catheter (up to 15 times on the treatment days and once the day after). One screening visit was planned up to 28 days before the start of treatment and one visit was planned about 7 days after the end of treatment.

The benefit-risk assessment was considered positive and justified the conduct of the planned study in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 55 years of age inclusive, at the time of signing the informed consent.
* Participants who were overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, body temperature, vital signs, and ECG.
* BMI within the range 18.0 to 29.9 kg/m^2 (inclusive) at the screening visit.
* Contraceptive used by men and female partners should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Exclusion Criteria:

* Known hypersensitivity to any study intervention (active substances or excipients of the preparations) to be used in the study - including e.g., non-investigational medicinal products, challenge agents, or rescue medication.
* Medical disorder, condition or history of such that would impair the participant's ability to take part in or complete this study in the opinion of the investigator.
* Diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study intervention(s) will not be normal.
* Use of systemic or topical medicines or substances which might influence the study objectives.
* Suspicion of drug or alcohol abuse.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-02 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Cmax for plasma finerenone concentration | 0-24 h post dose
  Cmax: maximum concentration.
AUC(0-tlast) for plasma finerenone concentration | 0-24 h post dose
  AUC = area under the curve, which was the total amount of finerenone in plasma

SECONDARY OUTCOMES:
Number of participants with treatment emergent adverse events (TEAEs) | After first administration of study intervention up to 3 days after end of treatment with study intervention
  AEs were considered to be treatment-emergent if they have started or worsened after administration up to 3 days after end of treatment with study intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Wuppertal GmbH, Wuppertal, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Click here to find further information and, after study completion, the study results according to Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/22292